CLINICAL TRIAL: NCT02095184
Title: GCC 1366: A Prospective Study of Neoadjuvant Non-Steroidal Aromatase Inhibitors to Evaluate Anti-Proliferative Response in Obese and Overweight Patients
Brief Title: GCC 1366: Anti-Proliferative Response to NeoAdjuvant AIs in Overweight and Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Suliat Nurudeen, Professor of Medicine, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00060250
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Postmenopausal; Hormone-Receptor Positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1: Normal Weight Anastrozole (Active Comparator): Cohort 1: Patients with BMI < 25.0 kg/m2 treated with anastrozole
  Interventions: Drug: Anastrozole
- Cohort 2: Overweight Anastrozole (Active Comparator): Cohort 2: Patients with BMI ≥ 25.0-29.9 kg/m2 treated with anastrozole
  Interventions: Drug: Anastrozole
- Cohort 3: Obese (Active Comparator): Cohort 3: Patients with BMI ≥ 30 kg/m2 treated with anastrozole
  Interventions: Drug: Anastrozole
- Cohort 4: Normal Weight Letrozole (Active Comparator): Cohort 4: Patients with BMI < 25.0 kg/m2 treating with letrozole
  Interventions: Drug: Letrozole
- Cohort 5: Overweight Letrozole (Active Comparator): Cohort 5: Patients with BMI ≥ 25.0-29.9 kg/m2 treating with letrozole
  Interventions: Drug: Letrozole
- Cohort 6: Obese Letrozole (Active Comparator): Cohort 6: Patients with BMI ≥ 30 kg/m2 treating with letrozole
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Anastrozole — 1 mg daily
  Other Names: Arimidex
  Arms: Cohort 1: Normal Weight Anastrozole; Cohort 2: Overweight Anastrozole; Cohort 3: Obese
Drug: Letrozole — 2.5 mg daily
  Other Names: Femara
  Arms: Cohort 4: Normal Weight Letrozole; Cohort 5: Overweight Letrozole; Cohort 6: Obese Letrozole

SUMMARY:
More than three quarter of patients with breast cancer are treated by hormone pills called tamoxifen and aromatase inhibitors (AIs). AIs are drugs that stop female hormone production. This hormone production mostly happens in fat, muscle, and breast tissue in postmenopausal women. The female hormone estrogen is an important hormone for the growth of breast cancer cells. Anastrozole (Arimidex®) and Letrozole (Femara®) are AIs that are approved by the Food and Drug Administration (FDA). They have been used since 2005 to treat women with early stage breast cancer.

When given before surgery (neoadjuvant), both anastrozole and letrozole have been shown to successfully shrink breast cancer tumors in most patients. In over 50% of patients, anastrozole and letrozole when given for about 4 months also helped to improve surgery outcomes. On top of that, whether or not a patient responds to anastrozole and letrozole before surgery can help the doctor decide whether that patient needs additional chemotherapy.

One of the things may influence the level of hormone is body weight. It has been previously shown that postmenopausal women with higher body fat have higher level of female hormone as well as an increased risk of breast cancer. This is likely due to an increase in aromatase activity in the fatty tissue. However, at the current time AIs are used at the same doses in all women with breast cancer no matter whether they have different body weight. Currently, we do not know for certain whether the same doses of AIs work as well in patients with higher body fat compared to patients with less body fat.

The purpose of this study is to see if women with higher body fat respond differently to AI treatment compared to women with lower body fat.

DETAILED DESCRIPTION:
GCC 1366 is a prospective randomized window trial to evaluate the anti-proliferative response in obese and overweight breast cancer patients treated with neoadjuvant non-steroidal aromatase inhibitors. Post-menopausal women over the age of 18 years with estrogen receptor positive Her 2 neu negative stage II-III breast cancer are eligible. Participants will be randomized according to BMI to neoadjuvant treatment with Arimidex or Letrozole.

A total of 90 patients will be enrolled with 15 patients in each cohort below.

* Cohort 1: Patients with BMI < 25.0 kg/m2 treating with anastrozole
* Cohort 2: Patients with BMI ≥ 25.0-29.9 kg/m2 treating with anastrozole
* Cohort 3: Patients with BMI ≥ 30 kg/m2 treating with anastrozole
* Cohort 4: Patients with BMI < 25.0 kg/m2 treating with letrozole
* Cohort 5: Patients with BMI ≥ 25.0-29.9 kg/m2 treating with letrozole
* Cohort 6: Patients with BMI ≥ 30 kg/m2 treating with letrozole

Based on the patients' calculated BMI, patients in each BMI category (normal, overweight, and obese) will be enrolled in the different cohorts as described above. The first 15 patients in each BMI category will be treated with anastrozole. After completion of enrollment in cohorts 1, 2, and 3, subsequent patients will be treated with letrozole in cohorts 4, 5, and 6.

Anastrozole 1 mg or Letrozole 2.5 mg oral daily will be administered and continued for a minimum of 14 days and a maximum of 28 days (2-4 weeks). Surgery will be performed between weeks 2-3 of treatment unless there are compelling medical or personal reasons that prevent a patient from having surgery during this time. In those cases, patients may continue anastrozole or letrozole up to 4 weeks before surgery. Surgery should be performed within 36 hours of the last dose of anastrozole or letrozole.

Tumor tissue that is obtained for diagnosis or to assess response to initial AI therapy will be utilized for correlative studies. A patient may be continued on anastrozole or letrozole beyond 4 weeks (up to 18 weeks) if in the opinion of the treating physician, the patient will benefit from extended endocrine therapy. In this context, patients will have a core needle biopsy performed at 2-4 weeks after treatment to assess Ki67 response to AI therapy. Patients with an appropriate response to treatment as determined by a decrease in Ki67 levels (≤10%) will be continued on AI treatment. Patients without an appropriate decrease in Ki67 levels will be recommended to have immediate surgery or a switch to neoadjuvant chemotherapy if desired by the patient and treating physician.

Patients on extended AI neoadjuvant treatment having core biopsy at 2-4 weeks for Ki67 determination for clinical decision making will be approached and consented for additional research tissues to be taken at the same time as the biopsy for Ki67 determination. Blood samples will be collected prior to starting treatment and within 3 days or on the day of surgery. Additional blood samples will be obtained as clinically necessary.

Clinical assessment will be performed prior to enrollment and within 3 days or on the day of surgery. For patients who continue neoadjuvant endocrine therapy past 4 weeks, clinical assessment will be performed at the time of clinical biopsy and every 4-6 weeks thereafter. For clinical evidence of progression, patients will be offered immediate surgery or switch to neoadjuvant chemotherapy at the discretion of the treating physician.

Radiological assessment including mammogram, ultrasound, and breast MRI will be performed as per standard of care.

Patients will be followed for 30 days on study after the last dose of anastrozole or letrozole prior to surgery. For patients who receive extended neoadjuvant therapy with anastrozole or letrozole and for patients who receive other primary treatment after anastrozole or letrozole administration prior to surgery, patients will be followed for 30 days on study after the last dose of anastrozole or letrozole. Patients continuing to experience adverse events attributable to anastrozole or letrozole will be followed as needed until resolution or stabilization of the adverse events. Patients who are either found to be ineligible or refuse to start treatment after consenting will not be followed and will be replaced. Their information will not be collected. After 30 days after the last dose of anastrozole or letrozole, if there are no continuing adverse events attributable to treatment, patients will be off study.

ELIGIBILITY:
Inclusion Criteria:

1. Female greater than or equal to 18 years.
2. Postmenopausal status, defined by no menstrual cycle for 12 months or surgical removal of ovaries.
3. Histologically confirmed adenocarcinoma of the breast.
4. Evidence of hormone sensitive, ER rich primary tumor defined by an Allred score of ≥6.
5. Human estrogen receptor -2 (HER2) negative in the primary tumor tissue as defined by:

   1. Grade 0 or 1+ staining intensity (on a scale of 0 to 3) by means of IHC analysis OR
   2. Grade 2+ staining intensity by means of immuno-histochemical (IHC) analysis with gene amplification on fluorescence in situ hybridization (FISH) < 2.0 OR
   3. Gene amplification on fluorescence in situ hybridization (FISH) < 2.0.
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3
7. Unresected operable breast cancer stage I-III with primary tumor ≥ 2.0 cm.
8. Ability to understand and the willingness to sign a written informed consent document.
9. Patients must not have received any prior chemotherapy, radiation therapy, or endocrine therapy for their current breast cancer. Patients who received tamoxifen or raloxifene or another agent for prevention of breast cancer may be included as long as the patient has discontinued the treatment at least one month prior to baseline study biopsy.
10. Patients must have an adequate tumor tissue sample prior to enrollment available for correlative studies as defined below: Core needle biopsy or incisional biopsy samples that can provide ≥ 5 unstained sections of 5 micron thickness. Fine needle aspiration (FNA) sample alone is not sufficient.
11. Patients must have adequate organ function as defined below:

    1. Total bilirubin within normal institutional limits
    2. aspartate aminotransferase (AST)(SGOT)/alanine aminotransferase (ALT)(SGPT) < 2.5 x institutional upper limit of normal
    3. Creatinine clearance ≥ 10 mL/min/1.73 m2

Exclusion Criteria:

1. Previous or current systemic malignancy within the past 3 years other than breast cancer or adequately treated cervical carcinoma in situ or basal/squamous carcinoma of the skin.
2. Patients may not be receiving any other investigational agent.
3. History of allergic reactions or hypersensitivity to compounds of similar chemical or biologic composition to anastrozole or letrozole.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Percent change in proliferative index (Ki67) after treatment with the standard dose anastrozole or letrozole in normal, obese, and overweight patients | 2-4 weeks Post-treatment
  Core biopsy

SECONDARY OUTCOMES:
To evaluate differences in baseline GP88 level | B,0-Prior to starting anastrozole or letrozole
  GP88-6ml Blood Serum Sample
To evaluate differences in baseline GP88 level | B,1-On the day of surgery or within 3 days of surgery
  GP88-6ml Blood Serum Sample
To evaluate differences in baseline GP88 level | B,2-obtained 2-4 weeks after initiation of AI therapy( for persons rec. extended neoadjuvant tx)
  GP88-6ml Blood Serum Sample
To assess estradiol levels at baseline and after treatment (in primary ER positive breast tumors) | Baseline
  10ml Blood Serum Sample
To assess estradiol levels at baseline and after treatment (in primary ER positive breast tumors) | 2-4 weeks Post treatment
  10ml Blood Serum Sample
To evaluate the association of AI-induced Ki67 response | Baseline
  (IHC)--Immunohistochemistry
To evaluate the association of AI-induced Ki67 response | 2-4 weeks Post-Treatment
  (IHC)--Immunohistochemistry
To evaluate differences in Oncotype Dx | Baseline(T0)
  Tumor Tissue Assay
To evaluate differences in Oncotype Dx | 2-4 Post-treatment
  Tumor Tissue Assay

OTHER OUTCOMES:
Metabolomic Profiling | B-0
  10ml Blood Serum Sample
Metabolomic Profiling | B-1
  10ml Blood Serum Sample
Metabolomic Profiling | B-2
  10ml Blood Serum Sample

CONTACTS AND LOCATIONS:
Overall Officials: Emily C Bellavance, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No